CLINICAL TRIAL: NCT04791423
Title: A Phase II/III, Randomized, Stratified, Observer-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Immunogenicity of GRAd-COV2 Vaccine in Adults Aged 18 Years and Older
Brief Title: Study of GRAd-COV2 for the Prevention of COVID-19 in Adults
Acronym: COVITAR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ReiThera Srl (Industry)
Collaborators: Istituto Nazionale per le Malattie Infettive "Lazzaro Spallanzani" IRCCS (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RT-CoV-2_01
Record Dates: First submitted 2021-02-22; First posted 2021-03-10 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2022-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: In the phase II part approximately 900 participants will be randomized in a 1:1:1 ratio to receive 1 single IM dose of GRAd-COV2 2x10^11 vp plus 1 dose of placebo after 21 days (n= approximately 300 subject) or 2 repeated (21 days apart) IM dose of GRAd-COV2 1x10^11 (n = approximately 300 subjects) or two doses of placebo (n = approximately 300 subjects) on day 1 and day 22.
  Once the phase III expansion is granted, according to the epidemic evolution,the availability on the market of alternative vaccine(s) and the characteristics of vaccination campaign, the phase III study design will be adapted following these 3 potential scenarios: 1) a superiority trial vs placebo on overall population; 2) a superiority trial vs placebo on an subset of population (low risk subjects for infection outcome) or 3) a non-inferiority trial vs the available alternative vaccine on a surrogate endpoint (correlates of protection), if available.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The phase II part of the study is a parallel-group preventive study with 3 arms that is participant and investigator blinded (observer blinded). The blinding of the phase III will depend on the scenario that will be implemented.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single dose of GRAd-COV2 (Experimental): 1 single IM dose of GRAd-COV2 2 x 10^11 vp plus 1 dose of saline placebo after 21 days
  Interventions: Biological: GRAd-COV2
- Double dose of GRAd-COV2 (Experimental): 2 repeated (21 days apart) IM dose of GRAd-COV2 1 x 10^11
  Interventions: Biological: GRAd-COV2
- Placebo (Placebo Comparator): Two doses of saline placebo on day 1 and day 22
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: GRAd-COV2 — GRAd-COV2 is a replication-defective gorilla adenoviral vector (GRAd) encoding the SARS-CoV-2 surface glycoprotein (S, Spike) antigen under the control of CMV immediate early promoter. The encoded Spike antigen is stabilized in pre-fusion conformation by introducing 2 proline residues
  Arms: Double dose of GRAd-COV2; Single dose of GRAd-COV2
Other: Placebo — Saline solution
  Arms: Placebo

SUMMARY:
Multicenter Study assessing the safety, efficacy, and immunogenicity of the candidate vaccine GRAd-COV2, compared to placebo, for the prevention of COVID-19. Participants will be adults ≥ 18 years of age who are healthy or have medically stable chronic diseases and are at increased risk for SARS-CoV-2 acquisition and COVID-19. In the phase II part approximately 900 participants will be randomized in a 1:1:1 ratio to receive i) 2 repeated (21 days apart) intramuscular (IM) doses of GRAd-COV2 at 1x10^11 viral particle (vp) (n = approximately 300 subjects) ii) 1 single IM dose of GRAd-COV2 at 2x10^11 vp plus 1 dose of placebo after 21 days (n= approximately 300 subject) or 2 doses of placebo (n = approximately 300 subjects) on day 1 and day 22. There will be 3 strata for randomization: ≥ 65 years, < 65 years and categorized to be at increased risk ("at risk") for the complications of COVID-19, and < 65 years "not at risk". Risk will be defined referring to the study participants' relevant past and current medical history. An independent Data Safety Monitoring Board will provide oversight, to ensure safe and ethical conduct of the Study; a Steering Committee will revise safety data (collected for 900 participants 1 week after dosing) and immunogenicity data (collected for 450 participants 5 weeks after the first dosing) generated in phase II part. Jointly DSMB and SC will recommend the expansion to phase III and the best regimen to be used.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female and male, ≥ 18 years of age at the time of consent
2. Medically stable such that, according to the judgment of the investigator, hospitalization within the study period is not anticipated and the participant appears likely to be able to remain on study through the end of protocol-specified follow-up. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months prior to enrollment
3. Able to understand and comply with study requirements/procedures based on the assessment of the investigator
4. Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
5. Female participants, (a) Women of childbearing potential must: Have a negative pregnancy test on the day of screening and on Day 1; use one highly effective form of birth control for at least 28 days prior to Day 1 and agree to continue using one highly effective form of birth control through 60 days following administration of study intervention.
6. Capable of giving signed informed consent.

Exclusion Criteria:

1. History of allergy to any component of the vaccine
2. History of Guillain-Barré syndrome or any other demyelinating condition
3. Significant infection or other acute illness, including fever > 37.3 °C on the day prior to or day of randomization
4. History of laboratory-confirmed SARS-CoV-2 infection
5. Any confirmed or suspected immunosuppressive or immunodeficient state, including asplenia (only for phase II)
6. Recurrent severe infections and use of immunosuppressant medication within the past 6 months
7. History of primary malignancy except for: (a) Malignancy with low potential risk for recurrence after curative treatment (for example, history of childhood leukaemia) or metastasis (for example, indolent prostate cancer) in the opinion of the site investigator. (b) Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease (c) Adequately treated uterine cervical carcinoma in situ without evidence of disease (d) Localized prostate cancer (only for phase II)
8. Clinically significant bleeding disorder (eg, factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following IM injections or vene puncture
9. Severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, and neurological illness, as judged by the Investigator (mild/moderate well-controlled comorbidities are allowed) (only for phase II)
10. Any other significant disease, disorder, or finding that may significantly increase the risk to the participant because of participation in the study, affect the ability of the participant to participate in the study, or impair interpretation of the study data
11. Receipt of, or planned receipt of investigational or licensed products indicated for the treatment or prevention of SARS-CoV-2 or COVID-19
12. Receipt of any vaccine (licensed or investigational) other than licensed influenza vaccines within 30 days prior to and after administration of study intervention
13. Receipt of immunoglobulins and/or any blood products within 3 months prior to administration of study intervention or expected receipt during the period of study follow-up
14. Involvement in the planning and/or conduct of this study (applies to both Sponsor staff and/or staff at the study site)
15. For women only - currently pregnant (confirmed with positive pregnancy test) or breast-feeding
16. Has donated ≥ 450 mL of blood products within 30 days prior to randomization or expects to donate blood within 90 days of administration of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10300 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with symptomatic laboratory confirmed COVID-19 | FROM > 28 DAYS POST FIRST DOSE (DAY 1) UP TO DAY 360
  A binary response, whereby a participant is defined as a COVID-19 case if their first case of SARS-CoV-2 RT-PCR-positive symptomatic illness occurs ≥ 28 days post first dose or ≥ 7 days after the second dose of study intervention (depending on the selected regimen).
Incidence of AEs, SAEs, MAAEs, and AESI | 28 DAYS POST EACH DOSE FOR AEs and FROM RANDOMIZATION UP TO DAY 360 FOR SAEs, MAAEs, and AESI
  1. Incidence of AEs for 28 days post each dose of study intervention.
  2. Incidence of SAEs, MAAEs, and AESIs from Day 1 post treatment through Day 360.
Incidence of local and systemic solicited AEs | 7 DAYS POST EACH DOSE OF STUDY INTERVENTION
  Incidence of local and systemic solicited AEs
Post-treatment GMTs in SARS-CoV2 S and/or RBD antibodies | from day 1 to day 36
  Post-treatment GMTs from day of dosing baseline value to 35 days post first dose in SARS-CoV-2 S and/or RBD antibodies.
Post-treatment GMFRs in SARS-CoV2 S and/or RBD antibodies | from day 1 to day 36
  Post-treatment GMFRs from day of dosing baseline value to 35 days post first dose in SARS-CoV-2 S and/or RBD antibodies.
Proportion of participants with post-treatment seroresponse (> 4-fold rise in titers) to the S and/or RBD antigens of GRAd-COV2 | from day 1 to day 36
  Proportion of participants with post-treatment seroresponse (> 4-fold rise in titers) to the S and/or RBD antigens of GRAd-COV2.

SECONDARY OUTCOMES:
Time to first SARS-CoV2 RT-PCR positive severe or critical symptomatic illness | FROM > 28 DAYS POST FIRST DOSE (DAY 1) UP TO DAY 360
  Time to first SARS-CoV-2 RT-PCR-positive severe or critical symptomatic illness occurring ≥ 28 days post first dose or ≥ 7 days after second dose of study intervention
Proportion of participants who have a post-treatment response for SARS-COV2 Nucleocapside antibodies | from Day 1 up to day 360
  Proportion of participants who have a post-treatment response (negative at baseline to positive post treatment with study intervention) for SARS-CoV-2 Nucleocapsid antibodies over time.
Time to first case of SARS-COV2 RT-PCR positive symptomatic illness using CDC criteria | FROM > 28 DAYS POST FIRST DOSE (DAY 1) UP TO DAY 360
  Time to first case of SARS-CoV-2 RT-PCR- positive symptomatic illness occurring ≥ 28 days post first dose or > 7 days after second dose of study intervention using CDC criteria.
Time to first COVID-19 related Emergency Department admission | FROM > 28 DAYS POST FIRST DOSE (DAY 1) UP TO DAY 360
  Time to first COVID-19-related Emergency Department admission occurring ≥ 28 days post single dose or ≥ 7 days post second dose of study intervention.
Time to COVID-19 related death | FROM > 28 DAYS POST FIRST DOSE (DAY 1) UP TO DAY 360
  Time to COVID-19 related death
Post-treatment GMTs in SARS-CoV-2 S and/or RBD antibodies | from day of dosing baseline value to 35 days after first dose
  Post-treatment GMTs from day of dosing baseline value to 35 days post first dose (14 days post second dose) in SARS-CoV-2 S and/or RBD antibodies
Post-treatment GMFRs in SARS-CoV-2 S and/or RBD antibodies | from day of dosing baseline value to 35 days after first dose
  Post-treatment GMFRs from day of dosing baseline value to 35 days post first dose (14 days post second dose) in SARS-CoV-2 S and/or RBD antibodies
Proportion of participants who have a post-treatment seroresponse (≥ 4-fold rise in titers) in S and/or RBD antigens of GRAd-COV2. | from day 1 to day 36
  The proportion of participants who have a post-treatment seroresponse (≥ 4-fold rise in titers from day of dosing baseline value to 35 days post first dose) to the S and/or RBD antigens of GRAd-COV2.
Post-treatment GMTs in SARS-CoV2 S neutralizing antibodies | from day of dosing baseline value to 35 days after first dose
  Post-treatment GMTs from day of dosing baseline value to 35 days post first dose (14 days post second dose) in SARS-CoV-2 neutralizing antibodies.
Post-treatment GMFRs in SARS-CoV2 S neutralizing antibodies | from day of dosing baseline value to 35 days after first dose
  Post-treatment GMFRs from day of dosing baseline value to 35 days post first dose (14 days post second dose) in SARS-CoV-2 neutralizing antibodies.
Proportion of participants with post-treatment seroresponse (> 4-fold rise in titers) in SARS-COV2 neutralizing antibodies | from day 1 to day 36
  Proportion of participants who have a post-treatment seroresponse (≥ 4-fold rise in titers from day of dosing baseline value to 35 days post first dose) to GRAd-COV2 as measured by SARS-CoV-2 neutralizing antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Lanini, Consultant, Principal Investigator — Istituto per le Malattie Infettive Lazzaro Spallanzani IRCCS
Locations (26):
- Italy (26):
  - Ospedale Vittorio Emanuele Ii, Bisceglie, Barletta- Andria-Trani
  - Istituto per le Malattie Infettive Lazzaro Spallanzani IRCCS, Roma, RM
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino
  - A.O. Sant'Anna E San Sebastiano Caserta, Caserta
  - Asst Di Cremona, Cremona
  - Azienda Ospedaliero-Universitaria Di Ferrara, Ferrara
  - Ao Ospedali Riuniti - Foggia, Foggia
  - E.O. Ospedali Galliera, Genova
  - Presidio Ospedaliero Nord-Ospedale Santa Maria Goretti Latina, Latina
  - Fondaz.Irccs Ca' Granda - Ospedale Maggiore Policlinico, Milan
  - Asst Fatebenefratelli Sacco, Milan
  - Ospedale S.Gerardo - Monza, Monza
  - Azienda Ospedaliera Dei Colli - P Cotugno, Napoli
  - Azienda Ospedaliera Universitaria Della Universita' Vanvitelli I Di Napoli, Napoli
  - Az.Osp.Univ.P.Giaccone, Palermo
  - Azienda Ospedaliero-Universitaria Di Parma, Parma
  - Policlinico S. Matteo - Pavia, Pavia
  - Azienda Usl Di Piacenza, Piacenza
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Azienda Ospedaliera Policlinico Umberto I, Roma
  - Policlinico A. Gemelli E C.I.C.- Policlinico Universitario A. Gemelli, Roma
  - Ospedale Amedeo Di Savoia, Torino
  - Azienda Sanitaria Universitaria Integrata Di Trieste, Trieste
  - Asst Dei Sette Laghi, Varese
  - Ospedale Unico Del Vercellese - Ospedale Sant'Andrea, Vercelli
  - Centro Ricerche Cliniche Di Verona Srl, Verona

REFERENCES:
- [Derived] Capone S, Fusco FM, Milleri S, Borre S, Carbonara S, Lo Caputo S, Leone S, Gori G, Maggi P, Cascio A, Lichtner M, Cauda R, Dal Zoppo S, Cossu MV, Gori A, Roda S, Confalonieri P, Bonora S, Missale G, Codeluppi M, Mezzaroma I, Capici S, Pontali E, Libanore M, Diani A, Lanini S, Battella S, Contino AM, Piano Mortari E, Genova F, Parente G, Dragonetti R, Colloca S, Visani L, Iannacone C, Carsetti R, Folgori A, Camerini R; COVITAR study group. GRAd-COV2 vaccine provides potent and durable humoral and cellular immunity to SARS-CoV-2 in randomized placebo-controlled phase 2 trial. Cell Rep Med. 2023 Jun 20;4(6):101084. doi: 10.1016/j.xcrm.2023.101084. Epub 2023 May 29. PMID 37315558